CLINICAL TRIAL: NCT02270450
Title: S1316, Prospective Comparative Effectiveness Trial for Malignant Bowel Obstruction
Brief Title: S1316, Surgery or Non-Surgical Management in Treating Patients With Intra-Abdominal Cancer and Bowel Obstruction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH); Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: S1316; U10CA037429 (NIH); 1R01HS021491-01A1 (AHRQ); S1316 (Other: SWOG); NCI-2014-01497 (Other: NCI)
Record Dates: First submitted 2014-10-10; First posted 2014-10-21 (Estimated); Results first posted 2022-11-21 (Actual); Last update posted 2023-03-30 (Actual); Status verified 2022-11

CONDITIONS: Constipation, Impaction, and Bowel Obstruction; Unspecified Adult Solid Tumor, Protocol Specific
MeSH Terms: conditions — Constipation; Intestinal Obstruction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Arm I (randomized to surgery) (Experimental): Patients undergo therapeutic conventional surgery (abdominal) as defined by the treating physician.
  Interventions: Procedure: therapeutic conventional surgery; Other: quality-of-life assessment
- Arm II (randomized to non-surgical management) (Experimental): Patients are offered gastrointestinal complications management/prevention (non-surgical management) as determined by the treating physician.
  Interventions: Procedure: gastrointestinal complications management/prevention; Other: quality-of-life assessment
- Arm III (no randomization, surgery) (Experimental): Patients undergo therapeutic conventional surgery (abdominal) as defined by the treating physician as in Arm I.
  Interventions: Procedure: therapeutic conventional surgery; Other: quality-of-life assessment
- Arm IV (no randomization, non-surgical management) (Experimental): Patients are offered gastrointestinal complications management/prevention (non-surgical management) as determined by the treating physician as in Arm II.
  Interventions: Procedure: gastrointestinal complications management/prevention; Other: quality-of-life assessment

INTERVENTIONS:
Procedure: therapeutic conventional surgery — Undergo abdominal surgery
  Arms: Arm I (randomized to surgery); Arm III (no randomization, surgery)
Procedure: gastrointestinal complications management/prevention — Undergo non-surgical management
  Other Names: complications management/prevention, gastrointestinal, management/prevention, gastrointestinal complications
  Arms: Arm II (randomized to non-surgical management); Arm IV (no randomization, non-surgical management)
Other: quality-of-life assessment — Ancillary studies
  Other Names: quality of life assessment

SUMMARY:
This partially randomized clinical trial studies surgery or non-surgical management in treating patients with intra-abdominal cancer and bowel obstruction. Bowel obstruction is a common problem for advanced cancer patients and can negatively affect quality of life. It is not yet known whether surgery or non-surgical management is the best treatment option for bowel obstruction and can lead to better quality of life.

DETAILED DESCRIPTION:
This partially randomized clinical trial studies surgery or non-surgical management in treating patients with intra-abdominal cancer and bowel obstruction. Bowel obstruction is a common problem for advanced cancer patients and can negatively affect quality of life. It is not yet known whether surgery or non-surgical management is the best treatment option for bowel obstruction and can lead to better quality of life.

ELIGIBILITY:
* Patient must have malignant bowel obstruction (MBO) as evidenced by all of the following:

  * Clinical evidence of a bowel obstruction (via history, physical, and radiographic examination)
  * Bowel obstruction below (distal to) ligament of Treitz
  * Intra-abdominal primary cancer with incurable disease
* Patients must have malignant bowel obstruction due to an intra-abdominal primary cancer (i.e. stomach, small bowel [including duodenum], pancreas, colon, rectum, appendiceal, ovarian, uterine, cervical, kidney, bladder, prostate, gastrointestinal stromal tumor [GIST] [all sites], and sarcoma)
* Patient must be able to tolerate a major surgical procedure based on clinical evaluation, status of their cancer, and any other underlying medical problems
* A member of the patient's surgical team must indicate equipoise for the benefit of the surgical treatment for MBO; the surgeon must respond "Yes" to each of the following questions and sign the S1316 Surgical Equipoise Documentation form for the patient to be eligible:

  * Is surgery for treatment of malignant bowel obstruction (MBO) being considered for this patient?
  * Do you have equipoise (If the treating team finds that an operation is required [e.g., for acute abdomen], or they would not offer the patient an operation [e.g., patient is too weak to tolerate surgery], then there is no equipoise)?
* Patients must not have signs of bowel perforation or "acute" abdomen as evidenced by free air on radiologic imaging or peritonitis on physical exam within 2 days prior to registration
* Patients must be registered to the study within 3 days after surgical consult for MBO and prior to any treatment (surgical or non-surgical) for MBO
* Patients must have Zubrod performance status of 0-2 within 7 days prior to registration
* Serum albumin must be planned to be collected after admission, but prior to treatment
* Patients must be able to complete the study questionnaires in English
* Patients or their legally authorized representative must be informed of the investigational nature of this study and must sign and give written informed consent in accordance with institutional and federal guidelines
* As a part of the Oncology Patient Enrollment Network (OPEN) registration process the treating institution's identity is provided in order to ensure that the current (within 365 days) date of institutional review board approval for this study has been entered in the system
* Patients must consent and provide both their contact information and that of their representative for a monthly 24-hour dietary recall phone call to be conducted by the Arizona Diet, Behavior and Quality of Life Assessment Lab

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 221 (Actual)
Dates: Start 2015-03-09 (Actual); Primary Completion 2021-04-01 (Actual); Study Completion 2021-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert S Krouse, M.D., F.A.C.S., Study Chair — University of Arizona
Locations (38):
- United States (34):
  - Cancer Center at Saint Joseph's, Phoenix, Arizona
  - Banner University Medical Center - Tucson, Tucson, Arizona
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Loma Linda University Medical Center, Loma Linda, California
  - Moffitt Cancer Center, Tampa, Florida
  - Rush University Medical Center, Chicago, Illinois
  - University of Kansas Cancer Center, Kansas City, Kansas
  - UMass Memorial Medical Center - University Campus, Worcester, Massachusetts
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Essentia Health Cancer Center, Duluth, Minnesota
  - Hackensack University Medical Center, Hackensack, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - South Shore University Hospital, Bay Shore, New York
  - North Shore University Hospital, Manhasset, New York
  - Long Island Jewish Medical Center, New Hyde Park, New York
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - University of Pennsylvania/Abramson Cancer Center, Philadelphia, Pennsylvania
  - Temple University Hospital, Philadelphia, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina
  - Methodist Le Bonheur Germantown Hospital, Germantown, Tennessee
  - The West Clinic - Wolf River, Germantown, Tennessee
  - Methodist Hospital, Memphis, Tennessee
  - University of Tennessee Health Science Center, Memphis, Tennessee
  - Baylor University Medical Center, Dallas, Texas
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - University Hospital, San Antonio, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Valley Health / Winchester Medical Center, Winchester, Virginia
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- University Health Network-Princess Margaret Hospital, Toronto, Ontario, Canada
- Instituto Nacional De Cancerologia, Bogotá, Colombia
- Instituto Nacional De Cancerologia de Mexico, Mexico City, Tlalpan, Mexico
- Instituto Nacional de Enfermedades Neoplasicas, Lima, Peru

REFERENCES:
- [Derived] Krouse RS, Anderson GL, Arnold KB, Thomson CA, Nfonsam VN, Al-Kasspooles MF, Walker JL, Sun V, Alvarez Secord A, Han ES, Leon-Takahashi AM, Isla-Ortiz D, Rodgers P, Hendren S, Sanchez Salcedo M, Laryea JA, Graybill WS, Flaherty DC, Mogal H, Miner TJ, Pimiento JM, Kitano M, Badgwell B, Whalen G, Lamont JP, Guevara OA, Senthil MS, Dewdney SB, Silberfein E, Wright JD, Friday B, Fahy B, Anantha Sathyanarayana S, O'Rourke M, Bakitas M, Sloan J, Grant M, Deutsch GB, Deneve JL. Surgical versus non-surgical management for patients with malignant bowel obstruction (S1316): a pragmatic comparative effectiveness trial. Lancet Gastroenterol Hepatol. 2023 Oct;8(10):908-918. doi: 10.1016/S2468-1253(23)00191-7. Epub 2023 Aug 1. PMID 37541263

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 221 patients were initially enrolled. 19 were ineligible: 12 with no small bowel obstruction, 3 with no confirmed bowel obstruction, 3 who were treated prior to registration and 1 with no intra-abdominal cancer. Another 3 patients were ineligible for analysis, due to withdrawal of consent prior to the end of their first hospitalization. In all, 199 patients were treated and evaluable for analysis: 49 randomized (24 surgery; 25 non-surgery) and 150 non-randomized (58 surgery; 92 non-surgery).
Period: Overall Study
Arm/Group | Arm I (Randomized to Surgery) | Arm II (Randomized to Non-surgical Management) | Arm III (no Randomization, Surgery) | Arm IV (no Randomization, Non-surgical Management)
Started | 24 | 25 | 58 | 92
Completed | 1 | 3 | 18 | 10
Not Completed | 23 | 22 | 40 | 82
Not completed — Refusal unrelated to adverse event | 3 | 1 | 5 | 14
Not completed — Progression/relapse | 1 | 2 | 4 | 9
Not completed — Death | 19 | 19 | 31 | 59

BASELINE CHARACTERISTICS:
Population: Eligible and evaluable participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (Randomized to Surgery) | Arm II (Randomized to Non-surgical Management) | Arm III (no Randomization, Surgery) | Arm IV (no Randomization, Non-surgical Management) | Total
Number analyzed (Participants) | 24 | 25 | 58 | 92 | 199
Age, Continuous [Median (Full Range); unit: years] | 63.4 [43.2 to 84.7] | 61.2 [45.7 to 82.3] | 61.1 [23.0 to 90.8] | 59.3 [32.7 to 85.6] | 60.4 [23.0 to 90.8]
Age, Customized [Count of Participants; unit: Participants]
  < 65 years | 13 | 17 | 36 | 65 | 131
  >= 65 years | 11 | 8 | 22 | 27 | 68
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 15 | 36 | 62 | 129
  Male | 8 | 10 | 22 | 30 | 70
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Race and ethnicity are categorized separately. Population: Race was not applicable for participants from Mexico and Peru.
  Participants
    Race - Black: number analyzed (Participants) | 16 | 20 | 58 | 92 | 186
    Race - Black | 6 | 7 | 13 | 16 | 42
    Race - White: number analyzed (Participants) | 16 | 20 | 58 | 92 | 186
    Race - White | 9 | 12 | 39 | 69 | 129
    Race - Other: number analyzed (Participants) | 16 | 20 | 58 | 92 | 186
    Race - Other | 1 | 1 | 1 | 3 | 6
    Race - Unknown: number analyzed (Participants) | 16 | 20 | 58 | 92 | 186
    Race - Unknown | 0 | 0 | 5 | 4 | 9
    Ethnicity - Hispanic | 9 | 5 | 6 | 13 | 33
    Ethnicity - Non-Hispanic | 14 | 18 | 51 | 78 | 161
    Ethnicity - Unknown | 1 | 2 | 1 | 1 | 5
Primary Cancer Site [Count of Participants; unit: Participants]
  Colorectal | 6 | 7 | 19 | 25 | 57
  Gynecologic | 10 | 12 | 14 | 38 | 74
  Other | 8 | 6 | 25 | 29 | 68
Body Mass Index (BMI), Continuous [Median (Full Range); unit: kg/m^2] | 23.8 [15.6 to 39.6] | 25.7 [16.4 to 37.9] | 24.4 [14.0 to 51.1] | 24.7 [16.0 to 50.4] | 24.6 [14.0 to 51.1]
Body Mass Index (BMI), Categorical [Count of Participants; unit: Participants]
  <18.5 (Underweight) | 3 | 2 | 7 | 6 | 18
  18.5 - <25 (Normal) | 10 | 10 | 26 | 45 | 91
  25 - <30 (Overweight) | 6 | 7 | 12 | 20 | 45
  >=30 (Obese) | 5 | 6 | 13 | 21 | 45
Albumin, Continuous [Mean (Standard Deviation); unit: g/dL] — Population: Number of participants analyzed differs from overall number of baseline participants due to missing data.
  g/dL
    number analyzed (Participants) | 24 | 25 | 58 | 91 | 198
    (all) | 3.1 (0.9) | 3.1 (0.7) | 3.2 (0.7) | 3.2 (0.7) | 3.2 (0.7)
Albumin, Child-Pugh [Count of Participants; unit: Participants]
  <2.8 | 7 | 7 | 18 | 25 | 57
  2.8 - 3.5 | 9 | 11 | 20 | 35 | 75
  >3.5 | 8 | 7 | 20 | 31 | 66
  Missing | 0 | 0 | 0 | 1 | 1
Ascites [Count of Participants; unit: Participants]
  No evidence | 8 | 12 | 26 | 43 | 89
  Evidence of ascites: trace/small amount | 11 | 7 | 24 | 29 | 71
  Evidence of ascites: large/massive amount | 5 | 6 | 8 | 20 | 39
Carcinomatosis [Count of Participants; unit: Participants]
  No evidence | 6 | 5 | 25 | 31 | 67
  Suspicion of carcinomatosis | 2 | 2 | 4 | 8 | 16
  Clear evidence: trace/small amount | 2 | 4 | 3 | 0 | 9
  Clear evidence: large/massive amount | 14 | 14 | 26 | 53 | 107
Performance Status [Count of Participants; unit: Participants] — Participants were graded according to the Zubrod Performance Status Scale:
  0 - Fully active, able to carry on all pre-disease performance without restriction.1 - Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light housework, office work. 2 - Ambulatory and capable of self-care but unable to carry out any work activities; up and about more than 50% of waking hours.
  Participants
    0 | 8 | 5 | 9 | 15 | 37
    1 | 6 | 9 | 29 | 50 | 94
    2 | 10 | 11 | 20 | 27 | 68
Number of Prior Malignant Bowel Obstructions (MBOs) [Count of Participants; unit: Participants]
  None | 17 | 16 | 32 | 51 | 116
  At least one | 5 | 4 | 21 | 31 | 61
  Unknown | 2 | 4 | 4 | 9 | 19
  Missing | 0 | 1 | 1 | 1 | 3
Care Providers [Count of Participants; unit: Participants] — Participants may have had more than one care provider.
  Participants
    Family member | 22 | 21 | 51 | 77 | 171
    Hospice/Skilled nursing | 1 | 1 | 0 | 6 | 8
    Other | 0 | 2 | 4 | 3 | 9
    No one | 1 | 2 | 5 | 11 | 19
Admitting Attending Physician Specialty [Count of Participants; unit: Participants] — "Medical Specialty" includes Family practice, Internal medicine, and Medical oncology.
  Participants
    Medical Specialty | 0 | 2 | 4 | 6 | 12
    General Surgery | 0 | 1 | 10 | 7 | 18
    Gynecologic Oncology | 3 | 4 | 5 | 30 | 42
    Surgical Oncology | 20 | 16 | 39 | 49 | 124
    Other | 1 | 2 | 0 | 0 | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Days Alive and Outside of the Hospital
Description: Number of days alive and outside of the hospital
Time Frame: From date of registration up to 91 days
Population: Eligible and evaluable participants
Measure: Mean (Standard Deviation); unit: days
Groups:
- Randomization Surgery: Patients who are randomized to surgical management undergo therapeutic conventional surgery (abdominal) as defined by the treating physician.
- Randomization Non-surgical Management: Patients who are randomized to non-surgical management are offered gastrointestinal complications management/prevention (non-surgical management) as determined by the treating physician.
- Patient Choice Surgery: Patients who choose surgical management undergo conventional surgery (abdominal) as defined by the treating physician as in Arm 1.
- Patient Choice Non-surgical Management: Patients who choose non-surgical management are offered gastrointestinal complications management/prevention (non-surgical management) as determined by the treating physician as in Arm 2.
Arm/Group | Randomization Surgery | Randomization Non-surgical Management | Patient Choice Surgery | Patient Choice Non-surgical Management
Number analyzed (Participants) | 24 | 25 | 58 | 92
days | 42.6 (32.2) | 43.9 (29.5) | 54.8 (27.0) | 52.7 (30.7)
Statistical Analysis 1: Comparison: Randomization Surgery vs Randomization Non-surgical Management vs Patient Choice Surgery vs Patient Choice Non-surgical Management; A linear regression model was applied to the combined data from the randomized and Patient Choice (non-randomized) pathways, using the intention to treat principle with a treatment indicator variable (surgical vs non-surgical management) based on assignment. The model compares the number of "good days" between patients assigned to surgery and patients assigned to non-surgical management; Test type: Superiority; p = 0.50, Regression, Linear — A p-value less than 0.05 is considered statistically significant; Adjusted for treatment, pathway, admitting attending physician specialty, Zubrod performance status, baseline albumin, and primary cancer site; Mean Difference (Net) = 2.87, Standard Error of Mean 4.3 — Comparing surgery to non-surgical management

2. Secondary Outcome: Number of Days in Hospital
Description: Length of initial hospital stay in days.
Time Frame: During initial hospitalization, from date of registration to a maximum of 53 weeks post registration
Population: Eligible and evaluable participants
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Randomization Surgery | Randomization Non-surgical Management | Patient Choice Surgery | Patient Choice Non-surgical Management
Number analyzed (Participants) | 24 | 25 | 58 | 92
days | 12.3 (9.3) | 12.8 (12.2) | 11.6 (7.8) | 6.2 (6.6)
Statistical Analysis 1: Comparison: Randomization Surgery vs Randomization Non-surgical Management vs Patient Choice Surgery vs Patient Choice Non-surgical Management; A linear regression model was applied to the combined data from the randomized and Patient Choice (non-randomized) pathways, using the intention to treat principle with a treatment indicator variable (surgical vs non-surgical management) based on assignment. The model compares the length of the initial hospital stay between patients assigned to surgery and patients and patients assigned to non-surgical management. An interaction term between treatment and pathway was included; Test type: Superiority; p = 0.64, Regression, Linear — For all secondary analyses, p-values should be interpreted cautiously as no adjustments for multiple comparisons were made; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = -1.09 — Comparing surgery to non-surgical management

3. Secondary Outcome: NG Tube Use
Description: Use of a nasogastric tube
Time Frame: During initial hospitalization, from date of registration to a maximum of 53 weeks post registration
Population: Eligible and evaluable participants
Measure: Count of Participants; unit: Participants
Arm/Group | Randomization Surgery | Randomization Non-surgical Management | Patient Choice Surgery | Patient Choice Non-surgical Management
Number analyzed (Participants) | 24 | 25 | 58 | 92
Participants
  Yes | 19 | 20 | 42 | 69
  No | 5 | 5 | 13 | 21
  Missing | 0 | 0 | 3 | 2
Statistical Analysis 1: Comparison: Randomization Surgery vs Randomization Non-surgical Management vs Patient Choice Surgery vs Patient Choice Non-surgical Management; A parallel logistic regression model was applied to the combined data from the randomized and Patient Choice (non-randomized) pathways, using the intention to treat principle with a treatment indicator variable (surgical vs non-surgical management) based on assignment. The model compares NG tube use vs no NG tube use between patients assigned to surgery and patients assigned to non-surgical management; Test type: Superiority; p = 0.60, Regression, Logistic — [p-value comment as in outcome 2, analysis 1]; [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 0.82 — Comparing surgery to non-surgical management

4. Secondary Outcome: Days of NG Tube Use
Description: Number of days a nasogastric tube was used during the patient's initial hospitalization
Time Frame: During entire initial hospitalization (admission to discharge) to a maximum of 53 weeks post registration
Population: Eligible and evaluable participants. Number of participants analyzed in the Patient Choice Surgery arm and Patient Choice Non-surgical Management arm differs from the overall number of eligible and evaluable participants due to missing data.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Randomization Surgery | Randomization Non-surgical Management | Patient Choice Surgery | Patient Choice Non-surgical Management
Number analyzed (Participants) | 24 | 25 | 55 | 90
days | 5.8 (4.1) | 7.7 (8.4) | 6.5 (5.6) | 5.1 (5.3)
Statistical Analysis 1: Comparison: Randomization Surgery vs Randomization Non-surgical Management vs Patient Choice Surgery vs Patient Choice Non-surgical Management; A linear regression model was applied to the combined data from the randomized and Patient Choice (non-randomized) pathways, using the intention to treat principle with a treatment indicator variable (surgical vs non-surgical management) based on assignment. The model compares the number of days of NG tube use between patients assigned to surgery and patients and patients assigned to non-surgical management; Test type: Superiority; p = 0.47, Regression, Linear — [p-value comment as in outcome 2, analysis 1]; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = 0.64 — Comparing surgery to non-surgical management

5. Secondary Outcome: MDASI-GI Symptom Assessment
Description: The MD Anderson Symptom Inventory for gastrointestinal cancer (MDASI-GI) was used to assess nausea, vomiting, pain, bloating, and constipation. The MDASI measures symptom severity on an 11-point scale, from 0 ("not present") to 10 ("as bad as you can imagine"). A difference of at least 1.2 points was considered a clinically meaningful difference between groups for MDASI-GI outcomes.
Time Frame: Assessed at 4 weeks post registration
Population: Eligible and evaluable participants who were alive with data at the time of the assessment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Randomization Surgery | Randomization Non-surgical Management | Patient Choice Surgery | Patient Choice Non-surgical Management
Number analyzed (Participants) | 11 | 11 | 31 | 41
score on a scale
  Nausea Severity | 0.64 (1.3) | 4.6 (3.8) | 1.9 (3.1) | 2.3 (3.0)
  Vomiting Severity | 0.64 (2.1) | 2.9 (3.5) | 0.58 (1.5) | 1.9 (3.0)
  Bloating Severity | 1.5 (2.3) | 3.9 (3.2) | 1.6 (2.4) | 2.3 (2.9)
  Pain Severity | 2.9 (3.1) | 5.7 (3.6) | 4.1 (3.3) | 3.8 (3.6)
  Constipation Severity | 0.55 (1.3) | 2.7 (3.9) | 0.77 (2.2) | 2.2 (3.4)
Statistical Analysis 1: Comparison: Randomization Surgery vs Randomization Non-surgical Management vs Patient Choice Surgery vs Patient Choice Non-surgical Management; A linear regression model was applied to the combined data from the randomized and Patient Choice (non-randomized) pathways, using the intention to treat principle with a treatment indicator variable (surgical vs non-surgical management) based on assignment. The model compares the MDASI-GI Symptom Assessment score for nausea severity between patients assigned to surgery and patients and patients assigned to non-surgical management. An interaction term between treatment and pathway was included; Test type: Superiority; p = 0.001, Regression, Linear — [p-value comment as in outcome 2, analysis 1]; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = -4.1 — Comparing surgery to non-surgical management
Statistical Analysis 2: Comparison: Randomization Surgery vs Randomization Non-surgical Management vs Patient Choice Surgery vs Patient Choice Non-surgical Management; A linear regression model was applied to the combined data from the randomized and Patient Choice (non-randomized) pathways, using the intention to treat principle with a treatment indicator variable (surgical vs non-surgical management) based on assignment. The model compares the MDASI-GI Symptom Assessment score for vomiting severity between patients assigned to surgery and patients and patients assigned to non-surgical management; Test type: Superiority; p = 0.008, Regression, Linear — [p-value comment as in outcome 2, analysis 1]; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = -1.63 — Comparing surgery to non-surgical management
Statistical Analysis 3: Comparison: Randomization Surgery vs Randomization Non-surgical Management vs Patient Choice Surgery vs Patient Choice Non-surgical Management; A linear regression model was applied to the combined data from the randomized and Patient Choice (non-randomized) pathways, using the intention to treat principle with a treatment indicator variable (surgical vs non-surgical management) based on assignment. The model compares the MDASI-GI Symptom Assessment score for bloating severity between patients assigned to surgery and patients and patients assigned to non-surgical management; Test type: Superiority; p = 0.04, Regression, Linear — [p-value comment as in outcome 2, analysis 1]; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = -1.31 — Comparing surgery to non-surgical management
Statistical Analysis 4: Comparison: Randomization Surgery vs Randomization Non-surgical Management vs Patient Choice Surgery vs Patient Choice Non-surgical Management; A linear regression model was applied to the combined data from the randomized and Patient Choice (non-randomized) pathways, using the intention to treat principle with a treatment indicator variable (surgical vs non-surgical management) based on assignment. The model compares the MDASI-GI Symptom Assessment score for pain severity between patients assigned to surgery and patients and patients assigned to non-surgical management. An interaction term between treatment and pathway was included; Test type: Superiority; p = 0.01, Regression, Linear — [p-value comment as in outcome 2, analysis 1]; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = -3.6 — Comparing surgery to non-surgical management
Statistical Analysis 5: Comparison: Randomization Surgery vs Randomization Non-surgical Management vs Patient Choice Surgery vs Patient Choice Non-surgical Management; A linear regression model was applied to the combined data from the randomized and Patient Choice (non-randomized) pathways, using the intention to treat principle with a treatment indicator variable (surgical vs non-surgical management) based on assignment. The model compares the MDASI-GI Symptom Assessment score for constipation severity between patients assigned to surgery and patients and patients assigned to non-surgical management; Test type: Superiority; p = 0.007, Regression, Linear — [p-value comment as in outcome 2, analysis 1]; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = -1.90 — Comparing surgery to non-surgical management

6. Secondary Outcome: Ability to Eat
Description: Ability to consume food was assessed based on self or caregiver-reported 24-hour dietary recalls. Dietary recalls were collected by trained assessors at the University of Arizona Cancer Center Behavioral Measurement and Interventions Shared Resource (BMISR) via telephone using standardized protocols and Nutrient Database for Research.
Time Frame: Assessed at 5 weeks post registration
Population: Eligible and evaluable participants who were alive with data at the assessment time
Measure: Count of Participants; unit: Participants
Arm/Group | Randomization Surgery | Randomization Non-surgical Management | Patient Choice Surgery | Patient Choice Non-surgical Management
Number analyzed (Participants) | 12 | 12 | 29 | 40
Participants
  Eating | 12 | 12 | 29 | 40
  Not eating | 0 | 0 | 6 | 7
Statistical Analysis 1: Comparison: Randomization Surgery vs Randomization Non-surgical Management vs Patient Choice Surgery vs Patient Choice Non-surgical Management; A parallel logistic regression model was applied to the combined data from the randomized and Patient Choice (non-randomized) pathways, using the intention to treat principle with a treatment indicator variable (surgical vs non-surgical management) based on assignment. The model compares ability to eat between patients assigned to surgery and patients and patients assigned to non-surgical management; Test type: Superiority; p = 0.52, Regression, Logistic — [p-value comment as in outcome 2, analysis 1]; Adjusted for treatment, admitting attending physician specialty, Zubrod performance status, baseline albumin, and primary cancer site; Odds Ratio (OR) = 0.64 — Comparing surgery to non-surgical management

7. Secondary Outcome: Overall Survival
Description: Time from date of registration to date of death due to any cause.
Time Frame: From date of registration to maximum of 53 weeks
Population: Eligible and evaluable participants
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Randomization Surgery | Randomization Non-surgical Management | Patient Choice Surgery | Patient Choice Non-surgical Management
Number analyzed (Participants) | 24 | 25 | 58 | 92
days | 86 [51 to 102] | 80 [39 to 102] | 156 [71 to 303] | 96 [71 to 144]
Statistical Analysis 1: Comparison: Randomization Surgery vs Randomization Non-surgical Management vs Patient Choice Surgery vs Patient Choice Non-surgical Management; A Cox proportional hazards regression model stratified by pathway (randomized vs Patient Choice) was used to estimate the effect of treatment assignment (surgery vs non-surgical management) on overall survival; Test type: Superiority; p = 0.12, Regression, Cox; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.70, 95% CI 2-sided [0.45 to 1.09] — Comparing surgery to non-surgical management

ADVERSE EVENTS:
Time Frame: From date of registration until death or 53 weeks post registration
Description: CTCAE Version 4.0 was used for routine toxicity reporting and Version 5.0 was used for Serious Adverse Event (SAE) reporting. Patients were assessed for AEs only while hospitalized. 199 patients were evaluable for AEs, including 24 on the Randomization Surgery arm, 25 on the Randomization Non-surgical Management arm, 58 on the Patient Choice Surgery arm, and 92 on the Patient Choice Non-surgical Management arm.
Groups:
- Randomization Non-surgical Management: Patients on the randomized to non-surgical management are offered gastrointestinal complications management/prevention (non-surgical management) as determined by the treating physician.
Arm/Group | Randomization Surgery | Randomization Non-surgical Management | Patient Choice Surgery | Patient Choice Non-surgical Management
All-Cause Mortality (participants affected / at risk) | 19/24 | 20/25 | 37/58 | 68/92
Serious Adverse Events (participants affected / at risk) | 2/24 | 3/25 | 5/58 | 16/92
Other Adverse Events (participants affected / at risk) | 5/24 | 1/25 | 12/58 | 14/92
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Randomization Surgery (N=24) | Randomization Non-surgical Management (N=25) | Patient Choice Surgery (N=58) | Patient Choice Non-surgical Management (N=92)
Anemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Cardiac arrest (Cardiac disorders) | 0 | 0 | 0 | 2
Death NOS (General disorders) | 0 | 2 | 0 | 2
Sepsis (Infections and infestations) | 0 | 0 | 0 | 4
Neoplasms benign, malignant and unspecified - Other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 5 | 10
Renal and urinary disorders-Other (Renal and urinary disorders) | 0 | 0 | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Randomization Surgery (N=24) | Randomization Non-surgical Management (N=25) | Patient Choice Surgery (N=58) | Patient Choice Non-surgical Management (N=92)
Anemia (Blood and lymphatic system disorders) | 4 | 1 | 8 | 13
Gastrointestinal fistula (Gastrointestinal disorders) | 3 | 0 | 3 | 0
Sepsis (Infections and infestations) | 2 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 2 | 0 | 2 | 2
Wound complication (Injury, poisoning and procedural complications) | 0 | 0 | 3 | 0
Wound dehiscence (Injury, poisoning and procedural complications) | 2 | 0 | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2019-06-18): https://cdn.clinicaltrials.gov/large-docs/50/NCT02270450/Prot_SAP_ICF_000.pdf